CLINICAL TRIAL: NCT03159130
Title: OnQ Pain Pump Effectiveness in Post Operative Pain Control in Bariatric Patients
Status: Withdrawn | Type: Observational
Why Stopped: PI dropped the study
Sponsor: William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 371884-1
Record Dates: First submitted 2017-05-12; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Morbid Obesity
Keywords: Pain pump catheters; bariatric surgery; OnQ pump; sleeve gastrectomy; continuous infusion catheter
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- receiving lidocaine: Each patient will receive an OnQ pain pump intra-operatively, with attachment to two OnQ catheters inserted on the lateral sides of the abdomen. Each catheter will be infused with 15 cc of 1% lidocaine.
- receiving injectable saline: Each patient will receive an OnQ pain pump intra-operatively, with attachment to two OnQ catheters inserted on the lateral sides of the abdomen. Each catheter will be infused with 15 cc of injectable saline.

SUMMARY:
This study will assess the efficacy of OnQ pain catheters in pain reduction in the bariatric surgical population and seeks to identify if a quantifiable improved post-operative course occurs in patients receiving a catheter filled with local anesthetic versus that achieved by patients who receive a catheter filled with injectable saline.

DETAILED DESCRIPTION:
This study will assess the efficacy of OnQ pain catheters in pain reduction in the bariatric surgical population. Approximately 12 to 15 weight reduction surgeries are performed at William Beaumont Army Medical Center each month. It is the current practice that each patient receiving the laparoscopic gastric sleeve or laparoscopic Roux-en-Y gastric bypass receive an OnQ pain catheter during the surgery to reduce post-operative pain. There have been limited studies to quantify the efficacy of these devices. This study will seek to identify if a quantifiable improved post-operative course occurs in patients receiving a catheter filled with local anesthetic versus that achieved by patients who receive a catheter filled with injectable saline.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Bariatric surgery
* Consents to be in protocol
* No local anesthetic allergy
* Will be having sleeve gastrectomy
* Doesn't have extensive scarring of abdominal wall that would prevent placement of OnQ catheter

Exclusion Criteria:

* declines to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a gastric sleeve procedure will be offered the opportunity to participate.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06 (Estimated); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Narcotic use | from admission to recovery room until discharge from the hospital (3-5 days)
  immediate post-operative narcotic use per patient

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Peirce, MD, Principal Investigator — William Beaumont Army Medical Center
Locations (1):
- William Beaumont Army Medical Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No